CLINICAL TRIAL: NCT07144696
Title: Study on the Improvement of Metabolic Indicators in Type 1 Diabetes Patients by Structured Education
Brief Title: Study on the Improvement of Metabolic Indicators in Type 1 Diabetes Patients
Acronym: T1D
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Peking University First Hospital (Other)
Responsible Party: Principal Investigator, Gu Nan, associate chief physician, Peking University First Hospital
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Supportive Care
Other Study IDs: 2024-447-002
Record Dates: First submitted 2025-08-04; First posted 2025-08-27 (Actual); Last update posted 2025-09-04 (Actual); Status verified 2025-08

CONDITIONS: Type 1 Diabetes Mellitus
MeSH Terms: conditions — Diabetes Mellitus, Type 1

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- structured education and regular follow-up (Experimental): education and regular follow-up
  Interventions: Behavioral: structured education and regular follow-up

INTERVENTIONS:
Behavioral: structured education and regular follow-up — Regularly carry out structured diabetes courses for patients with type 1 diabetes and offline teaching at Peking University First Hospital. On the basis of structured courses, regular outpatient follow-up visits will be conducted for patients, with on-site visits conducted at the Endocrinology Clinic of Peking University First Hospital. The usual visit period is once every 1-3 months, and the specific follow-up time nodes will be determined by medical staff based on the patient's condition. Each visit will last 1-3 hours, and each subject is expected to be followed up for 1 year. During each visit, collect the medical history and some personal information of the subjects, complete the routine physical examination, draw blood to test diabetes related indicators (including the determination of fasting

SUMMARY:
In this study, type 1 diabetes patients from the outpatient department of Peking University First Hospital were selected as the research objects. The investigators plan to recruit 150 participants. Using the course and teaching plan of "Take Control of My Life - Structured Education for Type 1 diabetes" issued by the China Type 1 diabetes Alliance, offline teaching is carried out regularly for type 1 diabetes patients, aiming to improve participants' knowledge and skills of disease self-management and improve participants' self-management behavior. The course content includes diabetes diet, exercise, blood glucose monitoring, insulin injection, complication prevention, psychological adjustment, etc. The training will take place at Peking University First Hospital. On the basis of structured courses, regular outpatient follow-up will be further carried out for patients to standardize their treatment behavior, improve their blood sugar compliance rate and delay the occurrence and development of diabetes complications. The subject visit is conducted on-site at the Endocrinology Clinic of Peking University First Hospital. The usual visit period is once every 1-3 months, and the specific follow-up time is determined by medical staff based on the subject's condition. Each visit lasts 1-3 hours, and each subject is expected to be followed up for 1 year. During each visit, collect the medical history and some personal information of the subjects, complete the routine physical examination, draw blood to test diabetes related indicators (including the determination of fasting and postprandial blood glucose, C-peptide, glycosylated hemoglobin, islet autoantibodies, blood lipids, liver and kidney functions), and screen diabetes complications. At the time of enrollment and after 1 year of follow-up, diabetes related questionnaires mainly related to diabetes self-management behavior and psychological emotions.

ELIGIBILITY:
Inclusion Criteria:

* ≥ 18 years old;
* It meets the WHO diagnostic criteria for diabetes and is diagnosed as type 1 diabetes;
* Capable and willing to participate in a 12 hour structured education course training;
* Capable and willing to accept regular outpatient follow-up visits;
* Voluntarily participate in this study and sign informed consent.

Exclusion Criteria:

* Non adult type 1 diabetes, type 2 diabetes and other special types of diabetes;
* Severe microvascular complications: proliferative retinopathy; Urinary albumin/creatinine>300mg/g, or 24-hour urinary protein quantification>1g/d; Uncontrolled painful diabetes neuropathy and significant diabetes autonomic neuropathy;
* Individuals who have undergone vascular intervention or amputation due to acute cerebrovascular accidents, acute coronary syndrome, or peripheral arterial disease requiring hospitalization within the first 3 months of selection;
* Blood pressure remains above 180/110mmHg and cannot be controlled within 160/110mmHg within one week;
* Blood creatinine clearance rate is less than 30ml/min/1.73m2 (calculated according to CKDEPI formula), alanine aminotransferase is ≥ 3 times the normal upper limit, total bilirubin is ≥ 2 times the normal upper limit and lasts for more than 1 week;
* Have used drugs that may affect blood sugar for more than one week within the past 12 weeks, such as oral/intravenous glucocorticoids, growth hormone, estrogen/progesterone, high-dose diuretics, antipsychotic drugs, etc; However, low-dose diuretics for blood pressure lowering purposes (hydrochlorothiazide<25mg/d, indapamide ≤ 1.5mg/d), as well as physiological doses of thyroid hormones used for replacement therapy, are not subject to this restriction;
* Systemic infection or severe accompanying diseases; Patients with malignant tumors or chronic diarrhea;
* Other situations that cause participants to be unable to cooperate in completing the study, such as severe cognitive impairment, mental illness, etc.
* The subject is uncooperative, unable to follow up, or the researcher determines that they may have difficulty completing the study.
* Other situations deemed unsuitable for inclusion by researchers. The research doctor will determine whether you are suitable to participate in this study based on your actual situation and the inclusion and exclusion criteria in the research plan.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 150 (Estimated)
Dates: Start 2025-08-05 (Actual); Primary Completion 2025-11-01 (Estimated); Study Completion 2026-08-31 (Estimated)

PRIMARY OUTCOMES:
Glycated hemoglobin | At baseline and 1-year follow-up
  Glycated hemoglobin between 4%~6% is normal

SECONDARY OUTCOMES:
self-management scale of type 1 diabetes for Chinese adults, SMOD-CA | At baseline and 1-year follow-up
  the minimum and maximum values is 0 and 120, and higher scores means better outcome
adjusted diabetes quality of life，A-DQOL | At baseline and 1-year follow-up
  the minimum and maximum values is 46 and 230, and higher scores means better outcome
Beck Depression Inventory, BDI | At baseline and 1-year follow-up
  the minimum and maximum values is 0 and 40, 0-5 points means healthy,6-15 points means mild depressive,16-25 points means has symptoms of depression,26-40 points means severe or severe depressive symptoms

CONTACTS AND LOCATIONS:
Locations (1):
- Peking University First Hospital, Beijing, China